CLINICAL TRIAL: NCT07105956
Title: Clinical Application of a Novel Radiolabeled Translocator Protein (TSPO) Targeted Small Molecular Probe in Neuroinflammation Imaging of Alzheimer's Disease.
Brief Title: Radiolabeled TSPO Targeted Molecular Probe in Alzheimer's Disease.
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250624-06-KS-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease (AD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the clinical application value of the novel radiolabeled TSPO-targeted molecular probe Gallium [68Ga]-DOTA-HK-011 in neuroinflammation imaging of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer for the trial, with the patient or their legal guardian signing the informed consent form.
* Volunteers are not limited by gender, and the age range is from 18 to 75 years old, including both ends.
* The patient is diagnosed with Alzheimer's disease (AD), supported by a positive amyloid PET scan.
* The patient has completed Tau PET scan.

Exclusion Criteria:

* Individuals with a history of allergy to drugs chemically or biologically similar to TSPO, a history of atopy, or currently suffering from allergic diseases.
* Use of anti-inflammatory drugs, including corticosteroids and immunosuppressants, within the past 14 days, which may interfere with the accuracy of inflammation imaging.
* Presence of other coexisting neurological diseases, such as stroke, Parkinson's disease, brain tumors, or mental disorders, including depressive disorder and schizophrenia.
* Severe cardiac, pulmonary, hepatic, or renal dysfunction, or uncontrolled systemic diseases; 5. Presence of metal implants contraindicated for MRI, including but not limited to cardiac pacemakers, artificial heart valves, and metal stents.
* Claustrophobia or inability to tolerate prolonged examinations.
* Pregnant women (defined as those with a positive urine pregnancy test) or breastfeeding women.
* Patients whose physical condition is unsuitable for radioactive tracer-based imaging examinations.
* Other circumstances deemed unsuitable for participation in the trial by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited through hospital electronic records and community health centers
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax of lesion uptake value | 60min after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jingasu, China